CLINICAL TRIAL: NCT06234345
Title: Randomized, Open-label, Parallel, Active-controlled, Multicenter Study of Efficacy and Safety of Fixed-dose Combination of Fluticasone /Formoterol /Glycopyrronium for the Treatment of Patients with Chronic Obstructive Pulmonary Disease
Brief Title: Study of Fluticasone/Formoterol/Glycopyrronium for the Treatment Chronic Obstructive Pulmonary Disease (TRIPLAR)
Acronym: TRIPLAR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF183
Record Dates: First submitted 2024-01-03; First posted 2024-01-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Formoterol Fumarate; Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: Experimental Group: Fluticasone Propionate 250 mcg/Formoterol Fumarate dihydrate 12 mcg/Glycopyrronium Bromide 25 mcg in the pharmaceutical form of hard capsule with powder for inhalation - 1 capsule per inhalation twice a day
  Comparator Group: Beclomethasone Dipropionate 100 mcg/Formoterol Fumarate dihydrate 6 mcg/Glycopyrronium Bromide 12.5 mcg in pharmaceutical form aerosol solution in pressurized metered dose device (pMDI) for inhalation (Trimbow® - Chiesi Farmacêutica Ltda.) - 2 triggering twice a day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluticasone Propionate 250 mcg/Formoterol Fumarate dihydrate 12 mcg/Glycopyrronium Bromide 25 mcg (Experimental): Fluticasone Propionate 250 mcg/Formoterol Fumarate dihydrate 12 mcg/Glycopyrronium Bromide 25 mcg in the pharmaceutical form of hard capsule with powder for inhalation - 1 capsule per inhalation twice a day
  Interventions: Drug: Fluticasone 250mcg/Formoterol 12mcg/Glycopyrronium 25mcg
- Trimbow® (Beclomethasone 100 mcg/Formoterol 6 mcg/Glycopyrronium 12.5 mcg) (Active Comparator): Beclomethasone Dipropionate 100 mcg/Formoterol Fumarate dihydrate 6 mcg/Glycopyrronium Bromide 12.5 mcg in pharmaceutical form aerosol solution in pressurized metered dose device (pMDI) for inhalation (Trimbow® - Chiesi Farmacêutica Ltda.) - 2 triggering twice a day
  Interventions: Drug: Comparator - Trimbow®

INTERVENTIONS:
Drug: Fluticasone 250mcg/Formoterol 12mcg/Glycopyrronium 25mcg — Participants randomized to this group will receive 1 capsule per inhalation twice a day
  Other Names: Fluticasone Propionate 250 mcg/Formoterol Fumarate dihydrate 12 mcg/Glycopyrronium Bromide 25 mcg
  Arms: Fluticasone Propionate 250 mcg/Formoterol Fumarate dihydrate 12 mcg/Glycopyrronium Bromide 25 mcg
Drug: Comparator - Trimbow® — Participants randomized to this group will receive 2 triggering twice a day
  Other Names: Trimbow® - Beclomethasone Dipropionate 100 mcg/Formoterol Fumarate dihydrate 6 mcg/Glycopyrronium Bromide 12.5 mcg
  Arms: Trimbow® (Beclomethasone 100 mcg/Formoterol 6 mcg/Glycopyrronium 12.5 mcg)

SUMMARY:
Several studies have demonstrated the benefits of the LAMA (Long-Acting Muscarinic Antagonists) + LABA (Long-Acting Beta-Agonists) + IC (inhaled corticosteroids) combination in the treatment of chronic obstructive pulmonary disease (COPD). The use of the triple combination in patients with severe airflow obstruction and a history of flares has been associated with improved lung function, improved patient-reported endpoints and prevention of flares, when compared to LABA, LABA + LAMA and LABA + IC. Furthermore, when compared to dual therapies LABA + IC and LABA + LAMA, triple therapy has been able to reduce all-cause deaths among chronic obstructive pulmonary disease (COPD) patients.

Previously published studies have demonstrated that the triple combination of Fluticasone 250 mcg/Formoterol 12 mcg/Glycopyrronium 12.5 mcg was able to improve lung function in chronic obstructive pulmonary disease (COPD) patients with a history of flares. There was also a significant improvement in the mMRC (modified-Medical Research Council) which began in the 2nd week of treatment and continued up to week 12. The association was considered safe and well tolerated, with only mild to moderate adverse events recorded in approximately 25% of the subjects treated in the study.

Furthermore, bioavailability studies performed with the components of the combination proposed as experimental drug - Fluticasone/Formoterol/Glycopyrronium - indicated that there is no pharmacokinetic interaction between the 3 active ingredients when they were administered concomitantly to healthy individuals under fasting conditions.

DETAILED DESCRIPTION:
This is a phase 3 non-inferiority, randomized, open-label study with active control to compare the efficacy and safety of a fixed-dose triple combination to another triple combination with already established efficacy in subjects with symptomatic chronic obstructive pulmonary disease (COPD).

This study will be conducted in two stages. Study Step 1 The primary assessment of non-inferiority will be performed after 12 weeks of treatment by assessing FEV1 (Forced expiratory volume in the first second) in relation to baseline.

Study Step 2 In a second step, it will be assessed whether the benefits of the new triple combination on respiratory symptoms and health-related quality of life are sustained in the long term and to determine the annual rate of flares in 52 weeks of treatment.

The study will comprise a screening phase, consisting of a screening and run-in visit lasting up to 14 days, and a treatment phase in which, after collecting baseline data (which includes assessment of FEV1 (Forced expiratory volume in the first second) and quality of life through a questionnaire), participants will be randomized and begin their respective treatments.

Visits during Step 1 of treatment will be performed at weeks 4 and 12. The week 12 visit will be the primary endpoint visit.

After 12 weeks, Step 2 of the study will begin with all participants who completed Step 1 and who agreed to remain in the study to receive Eurofarma's experimental drug for up to 52 weeks. Visits during this step will be performed at weeks 24, 36 and 52 to assess safety, quality of life, lung function and flare rate (exploratory endpoints).

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes who meet all of the following criteria will be included in the study:

  1. Signed Informed Consent Form (ICF).
  2. Male or female aged 40 or over.
  3. Medical diagnosis of chronic obstructive pulmonary disease (COPD) documented by post-bronchodilator FEV1/FVC (Forced Expiratory Volume in the 1st second/ Forced Vital Capacity) ratio < 0.7 (Previous examination report or examination performed at the screening visit).

Exclusion Criteria:

* Participants who meet any of the following criteria will be excluded from the study:

  1. Pregnant or lactating women.
  2. Current diagnosis of asthma without current diagnosis of chronic obstructive pulmonary disease (COPD). Observation: Subjects with a prior history of asthma are eligible if they have a current diagnosis of chronic obstructive pulmonary disease (COPD).
  3. Other respiratory disorders other than chronic obstructive pulmonary disease (COPD) (for example, but not restricted to: active tuberculosis, sarcoidosis, pulmonary fibrosis, pulmonary hypertension).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1252 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change to morning pre-dose FEV1 | week 12
  Change to morning pre-dose FEV1 at week 12 relative to baseline Forced expiratory volume in the first (FEV1).

SECONDARY OUTCOMES:
Change to SGRQ (Saint George's Respiratory Questionnaire) | week 12
  Change to SGRQ (Saint George's Respiratory Questionnaire) total score at week 12 compared to baseline
Change to the COPD (chronic obstructive pulmonary disease ) | weeks 4 and 12
  Change to the COPD (chronic obstructive pulmonary disease ) Assessment Test (CAT - questionnaire to measure the impact of COPD on a person's life) in weeks 4 and 12 in relation to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, Padrão, Brazil